CLINICAL TRIAL: NCT05115747
Title: Effect of Lower Body Positive Pressure Aerobic Training on Glycemic Indices and Quality of Life in Patients With Diabetic Polyneuropathy: Randomized Controlled Trial
Brief Title: Effect of Alter-G Training on Glycemic Control and Quality of Life in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Collaborators: King AbdulAziz City for Science and Technology (Other)
Responsible Party: Principal Investigator, Ashraf Abdelaal, ASSOCIATE PROFESSOR, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm AlQura Un
Record Dates: First submitted 2021-10-30; First posted 2021-11-10 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Polyneuropathy
Keywords: Diabetic neuropathy,Quality of Life,Blood Glucose,Hemoglobin
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: This interventional study aims to explore the effectiveness of the lower body positive pressure aerobic exercise training program on the glycemic control and the health-related quality of life in patients with diabetic polyneuropathy. Eighty eligible participants were randomly allocated to either group-A (0-percentage weight off-loading; 16-participants), group-B (25-percentage weight off-loading; 15-participants), group-C (50-percentage weight off-loading; 16-participants), group-D (75-percentage weight off-loading; 15-participants), and group-E (control group; 18-participants).
  Participants in the study groups received twelve-weeks mild to moderate intensity aerobic training program on the Alter-G anti-gravity treadmill.
  The Glycemic control (Fasting blood glucose in mg/dl, glycated hemoglobin, and health-related quality of life were evaluated at three time points: at the beginning of the study, after three months aerobic exercise training and three months post-training cessation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double: (Participants and outcome assessors).
  * Participants' random allocation was conducted by an independent person. The participants were unaware of the percentage of weight off-loading during the treadmill aerobic exercise training.
  * Outcomes Assessor kept blind about the group's allocation and the applied exercise training protocols.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- "Zero percentage" weight off-loading group-A (Experimental): This group received the Mild to moderate aerobic exercise training on the Alter-G treadmill with the full weight-bearing for three months.
  Interventions: Other: weight off-loading aerobic exercise training.
- "Twenty-five percentage" weight off-loading group-B (Experimental): This group received the Mild to moderate aerobic exercise training on the Alter-G treadmill with the twenty-five percentage" weight off-loading for three months.
  Interventions: Other: weight off-loading aerobic exercise training.
- "Fifty percentage" weight off-loading group-C (Experimental): This group received the Mild to moderate aerobic exercise training on the Alter-G treadmill with the fifty percentage" weight off-loading for three months.
  Interventions: Other: weight off-loading aerobic exercise training.
- "Seventy-five percentage" weight off-loading group-D (Experimental): This group received the Mild to moderate aerobic exercise training on the Alter-G treadmill with the seventy-five percentage" weight off-loading for three months.
  Interventions: Other: weight off-loading aerobic exercise training.
- Control group-E (No Intervention): Participated no aerobic exercise training.

INTERVENTIONS:
Other: weight off-loading aerobic exercise training. — Mild to moderate intensity weight off-loading aerobic exercise training on the anti-gravity Alter-G treadmill. (speed 8-12 mph, 50%-70% heart rate reserve "HRR", 12-16 score on the Borg's scale)
  Arms: "Fifty percentage" weight off-loading group-C; "Seventy-five percentage" weight off-loading group-D; "Twenty-five percentage" weight off-loading group-B; "Zero percentage" weight off-loading group-A

SUMMARY:
Aging is a natural process that is frequently accompanied by chronic physical or mental health problems. Aging as well as a sedentary lifestyle behavior may produce identical pathological and morphological changes. Saudi population, especially elderly people assume sedentary lifestyle, with little physical activity is a strong predisposition for developing a disability that adversely affects many aspects of physical and mental functions; mainly mobility and the ability to perform the basic daily living activities (ADL); resulting finally in increased risk of independence, loss of functionality, and falls. Type 2 diabetes mellitus (T2DM) is a widespread chronic metabolic disorder, accounts for 90-95% of all patients with diabetes. It is one of the most life-threatening public health challenges in the world, characterized by long term complications that almost involves all systems of the body. Polyneuropathy is the most common symptomatic complication in patients with type 2 diabetes mellitus, found in 50 to 60 % of patients over the age of sixty, with the impaired glycemic control and deteriorated quality of life are among the most debilitating problems in patients with diabetic polyneuropathy.

DETAILED DESCRIPTION:
Regular physical activity is an important component in healthy aging. Regular activity is very beneficial to our health as we age. Physical therapy can play an important role in the evaluation and treatment of older people with gait and balance disorders. Physical Therapy can help in the determination of the impairments produced by balance and gait abnormality and develop individualized plans aiming for identification of functional limitations.

Lower extremity aerobic exercise training (e.g., walking, treadmill and bicycle ergometer) is a good procedure to control and disrupt the progression of hyperglycemia in elderly with DPN. Furthermore; it improves lower limb muscle oxygen uptake, enhances the nerve conduction and proprioceptors sensitivity during activities. Lowe extremity aerobic exercise training can enhance balance, thereby reducing the falling risk. Aerobic exercise is also helpful in preventing age related lifestyle disease and improving quality of life (QOL) of the elderly. A conflict was clearly evoked between prescribing weight bearing and non- weight bearing exercise for elderly with diabetic polyneuropathy.

Weight bearing theoretical basis assumes that weight bearing activities such as walking are superior to other non- weight- bearing activities because of its ability to promote and restore muscular strength, joint proprioception and range of motion necessary to effectively perform typical daily activities. Although weight bearing training can significantly improve walking and balance abilities in patients with diabetic polyneuropathy compared with non- weight bearing training, but there were still not enough evidences to prove the ideal percentage level of weight reduction or unloading during practicing lower extremity training exercise in elderly with diabetic polyneuropathy. Quite recently, a new antigravity treadmill based on The National Aeronautics and Space Administration (NASA) technology was introduced. It permits low- load walking using an emerging technology called lower body positive pressure (LBPP) to modify body weight during ambulation. Few trials handled the utilization of LBPP technology and further trials are still warranted to to develop a more effective conservative and intervention treatment protocol for enhancing physical activities, quality of life and functional performance in elderly patients with diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diabetic polyneuropathy,
* Diagnosed as having uncontrolled type 2 diabetes mellitus, with glycosylated hemoglobin (HbA1c) value between 7 and 11 and fasting glucose level ranged from 7.0 -11.1 mmol/L,
* Age range from 60 and 80 years old,
* Established type 2 diabetes mellitus duration over 10 years, treated only with oral anti-diabetic agents (not taking insulin), treated only with Biguanide alone or (Sulfonylureas plus Biguanide) oral anti-diabetic drugs combination, with pharmacological treatment had to be stable for at least 3 months before the study,
* Cognitively competent and able to understand and follow instructions, capable of rationally interacting with others; understanding and answering the health related quality of life questionnaire (HRQL).

Exclusion Criteria:

* Type 1 DM, treated with insulin therapy or oral anti-diabetic therapy other than Biguanide alone or (Sulfonylureas plus Biguanide) combination,
* Younger than 60 or older than 80 years old,
* Patient with malnutrition (BMI < 21 kg/m2 or with recent weight loss > 5% body weight in the last month or > 10% in six months),
* Patients with established hypertension (resting systolic blood pressure > 140 mmHg and diastolic blood pressure > 90 mmHg,
* Active infection, drug abuse, participated in to an active rehabilitation program within last 6 months,
* With severe chronic or uncontrolled comorbid condition as recent myocardial infarction, unstable angina, acute congestive heart failure, third degree heart block and uncontrolled arrhythmia.
* With abnormal skin integrity e.g. wound or scares tissues or are on other complementary treatment,
* History of serious cerebrovascular or cardiovascular diseases, and severe debilitating musculoskeletal problems) that could interfere with the evaluation or treatment efficacy and patient safety or precluded the patient from attending and completing the treatment sessions.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Mean change in the fasting blood glucose level "in mg/dl" at three months. | Baseline and post-three months aerobic exercise training intervention, (at the 12th week)
  The fasting blood glucose (FBG) level "in mg/dl" will be evaluated in all participants at the baseline (at the beginning of the study) and at the end of the three-months Alter-G aerobic exercise training intervention (at the 12th week).
Mean change in the fasting blood glucose level in "mg/dl" at six months. | Baseline and after six months (three months post-training cessation; at the 24th week).
  The fasting blood glucose (FBG) level "in mg/dl" will be evaluated in all participants at the baseline (at the beginning of the study) and at the end of the six-months (three months post-training cessation).
Mean changes in the glycosylated hemoglobin level (HbA1c) at three months. | Baseline and post-three months aerobic exercise training intervention, (at the 12th week)
  The glycosylated hemoglobin level (HbA1c) will be evaluated in all participants at the baseline (at the beginning of the study) and at the end of the three-months Alter-G aerobic exercise training intervention (at the 12th week).
Mean changes in the glycosylated hemoglobin level (HbA1c) at six months. | Baseline and after six months (three months post-training cessation; at the 24th week).
  The glycosylated hemoglobin level (HbA1c) will be evaluated in all participants at the baseline (at the beginning of the study) and at the end of the six-months (three months post-training cessation).

SECONDARY OUTCOMES:
Mean changes in the health-related quality of life at three months. | Baseline and post-three months aerobic exercise training intervention, (at the 12th week)
  The health-related quality of life will be evaluated in all participants at the baseline (at the beginning of the study) and at the end of the three-months Alter-G aerobic exercise training intervention (at the 12th week).
Mean changes in the health-related quality of life at six months. | Baseline and after six months (three months post-training cessation; at the 24th week).
  The health-related quality of life will be evaluated in all participants at the baseline (at the beginning of the study) and at the end of the six-months (three months post-training cessation).

CONTACTS AND LOCATIONS:
Overall Officials: ASHRAF AM ABDELAAL, Principal Investigator — Umm Al-Qura University
Locations (1):
- Umm Al-Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No